CLINICAL TRIAL: NCT07372885
Title: A Multi-centre Phase I/II Trial of Granulocyte-augmented Cord Blood Transplantation for Young Adults With Very Poor Risk Acute Myeloid Leukaemia.
Brief Title: GRanulocyte Augmented Cord Blood Transplantation for Poor Risk leukaEmia
Acronym: GRACE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: King's College Hospital NHS Trust (Other); Institute of Cancer Research, United Kingdom (Other); The Christie NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mark Williams, Chief Investigator, University of Manchester
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 357519
Record Dates: First submitted 2025-11-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Stem Cell Transplantation; Stem Cell Transplantation, Hematopoietic; Cord Blood Stem Cell Transplantation; Cellular Therapy
Keywords: Grace; granulocyte-augmented cord blood transplantation; poor risk acute myeloid leukaemia; Cord Blood Transplantation; Myelodysplastic Syndrome; TP53; MECOM
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: This trial utilises an innovative early phase seamless design, integrating dose-escalation and randomised dose-optimisation which is built on latest FDA and MDICT guidance. Phase I (up to 30 patients) will include two components: dose-escalation and dose-optimisation to identify the Recommended Phase II Dose (RP2D). In the dose-escalation component, a modified 2-stage Bayesian Time-to-event Continual Reassessment Method (TITE-CRM) will be used to determine the maximum tolerated dose and tolerable doses among 4 dose schedules. In the dose optimisation, subsequent patients will be randomised to selected tolerable doses to determine final RP2D based on tolerability, activity and other key secondary endpoints in consultation with the integrated TSC/DMC. Phase II will assess preliminary efficacy at the RP2D, based on relapse free survival at 1 year using a single-stage Bayesian design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase I: T replete cord blood transplant + conditioning + 1 day Granulocytes (Active Comparator): All participants will receive a T replete cord blood transplant with a standardised conditioning regimen involving Fludarabine, Cyclophosphamide, Thiotepa, and TBI. A single pool of irradiated granulocytes will be given to participants for 1 day starting on the day of transplant.
  Interventions: Biological: Cord blood transplantation + conditioning + granulocytes of variable days according to study design
- Phase I: T replete cord blood transplant + conditioning + 3 day Granulocytes (Active Comparator): All participants will receive a T replete cord blood transplant with a standardised conditioning regimen involving Fludarabine, Cyclophosphamide, Thiotepa, and TBI. A single pool of irradiated granulocytes will be given daily to participants for 3 days starting on the day of transplant.
  Interventions: Biological: Cord blood transplantation + conditioning + granulocytes of variable days according to study design
- Active Comparator: Phase I: T replete cord blood transplant + conditioning + 5 day Granulocytes (Active Comparator): All participants will receive a T replete cord blood transplant with a standardised conditioning regimen involving Fludarabine, Cyclophosphamide, Thiotepa, and TBI. A single pool of irradiated granulocytes will be given daily to participants for 5 days starting on the day of transplant.
  Interventions: Biological: Cord blood transplantation + conditioning + granulocytes of variable days according to study design
- Active Comparator: Phase I: T replete cord blood transplant + conditioning + 7 day Granulocytes (Active Comparator): All participants will receive a T replete cord blood transplant with a standardised conditioning regimen involving Fludarabine, Cyclophosphamide, Thiotepa, and TBI. A single pool of irradiated granulocytes will be given daily to participants for 7 days starting on the day of transplant.
  Interventions: Biological: Cord blood transplantation + conditioning + granulocytes of variable days according to study design
- Phase II: T replete cord blood transplant + conditioning + Granulocytes at Recommended Phase II Dose (Experimental): All participants will receive a T replete cord blood transplant with a standardised conditioning regimen involving Fludarabine, Cyclophosphamide, Thiotepa, and TBI. A single pool of irradiated granulocytes will be given daily to all participants- at the Recommended Phase II Dose (RP2D)
  Interventions: Biological: Cord blood transplantation + conditioning + granulocytes of variable days according to study design

INTERVENTIONS:
Biological: Cord blood transplantation + conditioning + granulocytes of variable days according to study design — All participants will receive a T replete cord blood transplant with a standardised conditioning regimen involving Fludarabine, Cyclophosphamide, Thiotepa, and TBI. A single pool of irradiated granulocytes will be given daily to all participants- but for a variable number of days starting on the day of transplant according to study design (1,3,5 or 7 days). The study consists of two phases- Phase 1 has two components (dose escalation and dose optimisation) to identify the Recommended Phase II Dose (RP2D) of granulocytes. Phase 2 will assess preliminary efficacy based Relapse Free Survival at 1 year.

SUMMARY:
Allogeneic stem cell transplantation is the only potentially curative therapy for patients with high-risk Acute Myeloid Leukaemia, but relapse is common and remains the leading cause of death. Patients with certain mutations and those transplanted without first clearing their disease have very poor outcomes with most relapsing soon after transplant, and then surviving only a few months. A recent trial at the Royal Manchester Children's Hospital used cord blood stem cells alongside a type of white blood cell called 'granulocytes' and produced surprisingly good outcomes for children with very resistant leukaemia.

GRACE is a clinical trial for adults (<55 years) with Acute Myeloid Leukaemia that has not responded to chemotherapy or harbours mutations that predict a very poor response to conventional transplant. Participants will receive a transplant using umbilical cord blood and be given additional infusions of white blood cells, called granulocytes. The trial will be split into two parts:-The first will study the safety of this new approach. The experience of the investigators in children is that granulocyte infusions cause a fever, rash and expansion of another type of white blood cell called lymphocytes. Children that did not have this reaction did not respond to treatment. The investigators therefore believe that the reaction is necessary for the treatment to work, but the investigators must ensure that it is safe in adult patients. The trial design allows the investigators to determine the dose of granulocytes that is best tolerated and most likely to be effective.

The aim of the second part is to demonstrate that the new treatment is more effective than conventional transplantation.

The study will be conducted in three NHS transplant centres. Patients will be recruited over 36 months and followed up for a minimum of 1 year. The study is funded by Blood Cancer UK.

ELIGIBILITY:
1. Availability of a suitable cord blood unit
2. Age between 16 and 55 years
3. Primary diagnosis of Acute Myeloid Leukaemia (AML) or MDS/AML (as defined by ICC 2022) fitting one or more of the following criteria:

   * TP53 mutation (single- or multi-hit)
   * Presence of inv(3) (q21.3q26.2) or t(3;3)(q21.3;q26.2)
   * Adverse risk (as per ICC 2022) and >0.1% MRD by flow cytometry after 2 cycles of induction
   * AML (any risk) with partial remission (<10% blasts) after 2 cycles induction
   * Early relapse (<6 months) after chemotherapy alone (excluding t(16;16), inv(16) or t(8;21))
4. Bone marrow performed within 28 days of starting conditioning chemotherapy demonstrates either:

   * <10% blasts
   * >10% blasts with a hypocellular background (must be discussed with the trial team)
5. Suitable fitness and organ function as per the following criteria:

   * Glomerular filtration rate >50 mL/min/1.73m2
   * Ejection fraction >50%
   * FEV1 >65% without dyspnoea on mild activity
   * AST/ALT <3 x ULN
   * Bilirubin <1.5 x ULN (excluding Gilbert's syndrome)
   * Performance Status (ECOG) of 0 or 1
6. Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must agree to use appropriate, highly effective, contraception from the point of commencing therapy until 12 months after transplant

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity of Cytokine Release Syndrome (CRS) | Day 0 (day of allograft) to Day 28 post allograft
  Frequency and Severity of Cytokine Release Syndrome (CRS) assessed via ASTCT Consensus Grading for CRS
Frequency and Severity of Acute Graft vs Host Disease | Day 0 (day of allograft) to Day 100 post allograft
  Frequency and Severity of Acute Graft vs Host Disease assessed by modified Glucksberg criteria (revised by MAGIC)
Frequency and Severity of Chronic Graft vs Host Disease | Day 100 post allograft to Day 360 post allograft
  Frequency and Severity of Chronic Graft vs Host Disease assessed by NIH criteria
Frequency of Transplant Related Mortality (TRM) | Day 0 (day of allograft) to Day 100 post allograft
  Frequency of Transplant Related Mortality (TRM) defined as death due to any transplantation-related cause other than disease relapse
Frequency of Primary Graft Failure | Day 0 (day of allograft) to Day 28 post allograft
  Frequency of Primary Graft Failure
Rate of Relapse-Free Survival (RFS) | Day 0 (day of allograft) to Day 360 post allograft
  Relapse-free survival (RFS) rate: number of patients who remain relapse-free and alive within 1 year from transplant

SECONDARY OUTCOMES:
Frequency of Non-Relapse Mortality (NRM) | Day 0 (day of allograft) to Day 360 post allograft
  Non-relapse mortality (NRM): number of patients who die from aetiology not related to disease relapse.
Duration of Overall Survival | Day 0 (day of allograft) to Day 360 post allograft
  Overall survival: time from Day 0 to date of death from any cause. Patients who are alive will be censored at the date of last follow-up.
Duration of GvHD Free Relapse Free Survival (GRFS) | Day 0 (day of allograft) to Day 360 post allograft
  GvHD-free, relapse-free survival (GRFS): time from day to the first occurrence of any of the following events: acute grade III-IV and/or chronic GvHD requiring systemic immune suppressive treatment, disease relapse or progression, or death from any cause. Patients who are alive and free of any of these event will be censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Williams, BA MB BChir PhD MRCP FRCPath, Principal Investigator — University of Manchester; Mili N Shah, BSc MBBS MRCP FRCPath, Principal Investigator — Kings College Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - Kings College Hospital NHS Trust, London
  - The Royal Marsden Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT07372885/Prot_SAP_000.pdf